CLINICAL TRIAL: NCT00952861
Title: Antibiotic Treatment of Patients Admitted to Hospital With Acute Exacerbation of COPD. Effect of 1 Day of Antibiotic Therapy Compared to 6 Days of Therapy in Patients Who Are Stable After 24 Hours
Brief Title: Antibiotics in Chronic Obstructive Pulmonary Disease (COPD)
Acronym: TAExaCOP
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Stopped due to poor recruitment
Sponsor: Odense University Hospital (Other)
Collaborators: Kolding Sygehus (Other); Svendborg Hospital (Other); Fredericia Hospital (Unknown); Naestved Hospital (Other); Hillerod Hospital, Denmark (Other); Region Syddanmark (Other); Danmarks Lungeforening (Other); Danish National Research Foundation (Other)
Responsible Party: Court Pedersen / professor, Department of Infectious Diseases, Odense University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OUH-INF-1
Record Dates: First submitted 2009-07-24; First posted 2009-08-06 (Estimated); Last update posted 2010-08-11 (Estimated); Status verified 2010-06

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Chronic obstructive pulmonary disease; Infection; Antibiotics
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Infections | interventions — Doxycycline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Doxycycline (Active Comparator): Doxycycline 200 mg QD in 5 days
  Interventions: Drug: Doxycycline
- Placebo (Placebo Comparator): Matching placebo QD i 5 days
  Interventions: Drug: Placebo (matching)

INTERVENTIONS:
Drug: Doxycycline — 200 mg QD in 5 days
  Arms: Doxycycline
Drug: Placebo (matching) — Placebo QD i 5 days
  Arms: Placebo

SUMMARY:
It is not clear whether antibiotic therapy is needed in patients with mild to moderate exacerbation of chronic obstructive lung disease. The aim of the study is to compare the effect of 1 day of treatment with 6 days of treatment in patients who are admitted to hospital and being clinical stable (as judged by their physician) 24 hours after hospitalization

ELIGIBILITY:
Inclusion Criteria:

* Age above 50 years
* History of smoking
* History of COPD
* Antibiotics for 24 hours
* At least 2 of the following: dyspnoea, coughing with sputum, and sputum with purulence
* Informed consent

Exclusion Criteria:

* Pneumonia
* Antibiotics for more than 36 hours
* Antibiotics for other infection
* Prednisolone, more than 0.5 mg/kg body weight/24 hours for more than 3 days
* Malignancy
* Other pulmonary disease
* Immune deficiency
* Not able to tolerate doxycycline
* Severe heart, liver or kidney disease
* Epilepsia
* Not stable 24 hours after hospital admission
* Need for assisted ventilation

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2009-10; Primary Completion 2010-10 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
6 minutes walking distance | Day 14

SECONDARY OUTCOMES:
Time to next episode of acute exacerbation | Days 14, 30, 90 and 180

CONTACTS AND LOCATIONS:
Overall Officials: Court Pedersen, MD, Study Chair — Odense University Hospital
Locations (1):
- Odense University Hospital, Odense, Denmark